CLINICAL TRIAL: NCT05033119
Title: PROSA: Prolactin, Sex Hormones, Growth and Metabolic Biomarkers in Children and Adolescents on Antipsychotics
Acronym: PROSA
Status: Active, not recruiting | Type: Observational
Sponsor: Ulla Schierup Nielsen (Other)
Collaborators: North Denmark Region (Other Government); Central Denmark Region (Other); Mental Health Centre Copenhagen, Bispebjerg and Frederiksberg Hospital (Other)
Responsible Party: Sponsor-Investigator, Ulla Schierup Nielsen, National Coordinating Principal Investigator, Aalborg Psychiatric Hospital
Organization: Aalborg University Hospital (Other)
Other Study IDs: N-20210029
Record Dates: First submitted 2021-08-27; First posted 2021-09-02 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Hyperprolactinemia; Puberty Disorders; Metabolic Syndrome; Growth Disorders; Antipsychotics and Neuroleptics Toxicity
MeSH Terms: conditions — Hyperprolactinemia; Metabolic Syndrome; Growth Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objectives of this study are:

1. To determine the prevalence and degree of hyperprolactinemia in children and adolescents aged 7-18 years receiving antipsychotic medications
2. To determine the associations between serum-prolactin and sex hormones / metabolic biomarkers/ clinical symptoms in this population. If clinically relevant associations are found: To determine a potentially existing "no harm" serum-prolactin threshold
3. To determine associations between previous cumulative prolactin-exposure and current pubertal development / growth

ELIGIBILITY:
Inclusion Criteria:

* • In daily treatment with antipsychotic medication belonging to Anatomical Therapeutic Chemical (ATC) group N05A (except N05AN lithium) for a minimum duration of 3 months prior to inclusion

Exclusion Criteria:

* Eating Disorder
* Medical treatment to change sex
* Pregnancy or lactation

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All outpatients aged 7-18 years receiving treatment with antipsychotics at the Department of Child and Adolescent Psychiatry, Aalborg University Hospital, the Department of Child and Adolescent Psychiatry, Aarhus University Hospital and at the Child and Adolescent Mental Health Center, Copenhagen University Hospital, Capital Region will be invited to participate in the study.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Prevalence of hyperprolactinemia | 2 years

SECONDARY OUTCOMES:
associations between serum-prolactin and sex hormones / metabolic biomarkers / clinical symptoms | 2 years
associations between previous prolactin-exposure and current pubertal development / growth | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ulla S Nielsen, Study Director — Research Unit for Child and Adolescent Psychiatry, Aalborg,
Locations (3):
- Denmark (3):
  - Research Unit for Child and Adolescent Psychiatry, Aalborg University Hospital, Denmark, Aalborg
  - Aarhus University Hospital, Aarhus
  - Child and Adolescent Mental Health Center Capital Region, Denmark, Copenhagen

IPD SHARING:
Plan to Share IPD: No